CLINICAL TRIAL: NCT02886572
Title: Outcome in Patients With 4 or More Brain Metastases Treated With Single-Isocenter, Multi-Target (SIMT) Stereotactic Radiosurgery: A Prospective Single-arm Study in Adults With Brain Metastases
Brief Title: SIMT Stereotactic Radiosurgery Outcomes Study
Acronym: SIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00075429
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Radiosurgery (Experimental): All subjects will receive stereotactic radiosurgery(SRS) following the RTOG Stereotactic Radiotherapy Guidelines available at http://dx.doi.org/10.1016/j.prro.2011.06.014
  Interventions: Radiation: Stereotactic radiosurgery

INTERVENTIONS:
Radiation: Stereotactic radiosurgery — Linear-accelerator-based, single-isocenter, image-guided stereotactic radiosurgery
  Other Names: SRS

SUMMARY:
The purpose of this study is to determine the effectiveness and efficiency of Single Isocenter Multi-target Stereotactic Radiosurgery (SIMT SRS) in patients with four or more brain metastases

DETAILED DESCRIPTION:
Forty patients with four or more brain metastases will be enrolled prior to radiosurgery. A planning MRI brain scan will be performed with GD-DPTA within one week prior to radiosurgery, per the standard of care. Neurocognitive (Mini-Mental Status Examination (MMSE), Trail-making test A&B, Hopkins Learning Verbal (HVLT)) and functional assessment of cancer therapy-brain (FACT- Br) will be obtained prior to radiosurgery. Dose will be prescribed to the maximum isodose line encompassing the resulting PTV using the dose guidelines as described below.

The primary endpoint will be the proportion of patients who live longer than predicted based on the diagnosis-specific GPA score. The Kaplan-Meier estimator will be used to describe the survival of all patients treated with SIMT SRS. Secondary endpoints will be the rate of recurrence at the treated metastases sites, the rate of new brain metastases at a site different from the SRS-treated metastases sites, the rate of death due to neurological causes, and the prevalence of significant adverse events. Exploratory endpoints include change over time in neurocognition and quality of life, quantification of dosimetric measures, the rate of salvage therapy, the rate of radionecrosis at the SRS treatment sites, and the rate and intensity of steroid-usage post-SRS.

All patients will be evaluated for neurocognitive function via MMSE, HVLT, and Trail-making tests A & B, quality of life via FACT-Br, and for local recurrence via MRI every 3 months over the course of the study. These evaluations will be done at regular follow-up evaluations or when local recurrence is suspected on the basis of symptoms. Distant recurrence is defined as the appearance of new brain metastases at a site different from that of the original metastases. Recurrence will further be defined as a new area of enhancement that measures greater than 5 millimeters in the axial plane on MRI. The length of time to recurrence of the original brain metastases will be calculated from the date of the brain metastases radiosurgery to the date that a recurrence was detected by MRI. Patients with suspected recurrent tumor and/or who are symptomatic may undergo a stereotactic biopsy to evaluate for radionecrosis versus recurrent brain metastases, as is standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. A contrast-enhanced MRI scan showing = or > 4 brain metastases.
2. Age >/=18 years of age.
3. KPS >/= 70
4. Patient must have a graded prosnostic score (GPA) score 0.5 or greater
5. Life expectancy of at least 3 months
6. Postoperative patients with resected brain metastases are eligible.
7. Largest lesion < 4cm diameter
8. Must be a candidate for MRI imaging
9. Previous cranial stereotactic radiosurgery (SRS) or whole brain radiation therapy (WBRT) is allowed if > 3 months prior to SIMT
10. Must be capable of providing informed consent

Exclusion Criteria:

1. Primary lesion with radiosensitive histology (i.e., small cell carcinoma, germ-cell tumors, lymphoma, leukemia, and multiple myeloma).
2. Metastases within 2 mm of the optic apparatus
3. Patients unable to obtain MRI
4. Evidence of leptomeningeal disease
5. Greater than 10 brain metastases
6. Pregnant women are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace J. Kim, MD PhD, Principal Investigator — Duke University Medical Center, Radiation Onoclogy
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim GJ, Buckley ED, Herndon JE, Allen KJ, Dale TS, Adamson JD, Lay L, Giles WM, Rodrigues AE, Wang Z, Kelsey CR, Torok JA Jr, Chino JP, Fecci PE, Sampson JH, Anders CK, Floyd SR, Yin FF, Kirkpatrick JP. Outcomes in Patients With 4 to 10 Brain Metastases Treated With Dose-Adapted Single-Isocenter Multitarget Stereotactic Radiosurgery: A Prospective Study. Adv Radiat Oncol. 2021 Jul 23;6(6):100760. doi: 10.1016/j.adro.2021.100760. eCollection 2021 Nov-Dec. PMID 34934856

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Radiosurgery
Started | 40
Survival Analysis Population (All subjects were included in the survival analysis including 8 subjects who died prior to the first MRI.) | 40
Distant Brain Recurrence | 32
Local Recurrence | 32
Time to Neurologic Death | 32
SRS Related Adverse Events | 32
Completed | 32
Not Completed | 8
Not completed — Death | 8

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Karnofsky performance status [Median (Full Range); unit: units on a scale (percentage)] — The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment. The lower the Karnofsky score (presented as a percentage), the worse the survival for most serious illnesses. The score ranges from 0 (dead) to 100 (normal, no evidence of disease).
  units on a scale (percentage) | 90 [70 to 100]
Number of Metastases per participant [Median (Full Range); unit: metastases] | 6 [4 to 10]
Prior brain surgery for metastasis [Count of Participants; unit: Participants] | 36
Prior stereotactic radiosurgery or whole brain radiation [Count of Participants; unit: Participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Live Longer Than Predicted According to the Graded Prognostic Assessment (GPA) Score
Description: Calculated from the time of protocol Stereotactic RadioSurgery (SRS). The GPA incorporates four factors: age, KPS (Karnofsky Performance Score), ECM (extracranial metastases) and number of BM (brain metastases). Each factor is given a score of 0, 0.5 or 1.0 and GPA is calculated as a sum score of all four factors. The GPA has four groups: the GPA 0-1 with median survival of 2.6 months; GPA 1.5-2.5 with survival of 3.8 months; GPA 3 with median survival of 6.9 months and GPA 3.5-4.0 with the best median survival of 11 months.
Time Frame: Up to 24 months after SRS
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 32
Participants | 22

2. Secondary Outcome: Number of Participants Who Experience Local Brain Recurrence Within 1 Year of SIMT SRS Treatment
Description: Local recurrence of brain metastases is based on serial MRIs every 3 months and estimated by Kaplan-Meier analysis.
Time Frame: Up to 12 months after SRS
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 32
Participants | 4

3. Secondary Outcome: Number of Participants Who Are Dead Within 1 Year of SIMT SRS Treatment Due to Neurologic Reasons
Description: Time to neurologic death is defined as the time between initiation of SIMT SRS and death due to neurologic causes and is estimated using Kaplan-Meier analysis.
Time Frame: Up to 12 months after SRS
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 40
Participants | 30

4. Secondary Outcome: Number of Participants Who Experience a New Brain Metastasis at a Site Different From the Original Brain Metastasis Site 1 Year After SIMT SRS Treatment
Description: Distant recurrence of brain metastases is based on serial MRIs every 3 months and estimated by Kaplan-Meier analysis.
Time Frame: Up to 12 months after SRS
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 40
Participants | 19

5. Secondary Outcome: Number of Participants Who Experience Grade 3, 4, or 5 Neurologic Adverse Events Attributable to SIMT SRS
Description: Adverse Events only included those that were deemed by the PI to be related to the SIMT SRS treatment.
Time Frame: Up to 12 months after SRS
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 32
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Serious Adverse Events were only collected if they were grade 3, 4, or 5 event and were deemed by the Principal Investigator to be probably, possibly, or definitely related to the SRS treatment.
Arm/Group | Stereotactic Radiosurgery
All-Cause Mortality (participants affected / at risk) | 39/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 16/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Radiosurgery (N=40)
Eye disorders: other, specify (decrease visual acuity) (Eye disorders) | 2 (2)
Nausa (Gastrointestinal disorders) | 10 (10)
Vomiting (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 16 (16)
Gait disturbance (General disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Scalp pain (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT02886572/Prot_SAP_000.pdf